CLINICAL TRIAL: NCT07013266
Title: Burnout Syndrome Among Anesthesiologists in Turkey: A Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selcan Akesen, Associate Professor, Uludag University
Other Study IDs: 2025-2/14
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Burnout, Professional; Burnout, Psychological
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Burnout syndrome is a condition in which an individual experiences loss of self-esteem, chronic fatigue, feelings of helplessness, and hopelessness in their professional work life and human relationships. This study aims to evaluate the prevalence of burnout syndrome among anesthesiologists working in Turkey, analyze the potential causes and adverse consequences of this syndrome's increase, and provide recommendations for its reduction.

ELIGIBILITY:
Inclusion Criteria:

I. Agreed to participate by completing the online survey form. II. Proficient in the Turkish language. III. Anesthesiology and Reanimation specialists currently practicing in the Republic of Turkey.

Exclusion Criteria:

I. Users who do not provide consent to share the requested information in the survey form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anesthesiology and Reanimation specialists currently practicing in the Republic of Turkey.
  All anesthesiology and reanimation specialists registered with the Turkish Society of Anesthesiology and Reanimation will be contacted via email through the society. An online survey link will be provided to participants within this email. Participants who agree to take part in the survey and meet the inclusion criteria will be included in the study, and their responses to the questions will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Burnout Syndrome as measured by the Maslach Burnout Inventory | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Selcan Akesen, Principal Investigator — Uludağ Üniversitesi

IPD SHARING:
Plan to Share IPD: No